CLINICAL TRIAL: NCT06669117
Title: A First-In-Human (FIH) Phase I/II Open-label, Multicentre, Dose Escalation and Expansion Trial of VERT-002 in Patients With Locally Advanced or Metastatic Solid Tumors Including Non-small Cell Lung Cancer (NSCLC) Harboring Mesenchymal-Epithelial Transition (MET) Alterations
Brief Title: FIH Trial of VERT-002 in Patients With Locally Advanced or Metastatic Solid Tumors With MET Alterations
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: F60089IV101; 2024-512760-64-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-24; First posted 2024-11-01 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Solid Tumor; MET Alteration
Keywords: Locally advanced or metastatic solid tumors; MET alteration; Non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- VERT-002 (PFL-002) (Experimental): Part 1: Dose escalation (Phase Ia): VERT-002 will be administered via intravenous (IV) infusion every 2 weeks. 4 provisional doses are planned. An alternative regimen may be tested informed by the emerging data
  Part 2a: Preliminary Activity Assessment (Phase Ib): One dose & schedule selected from Part 1
  Part 2b: Dose range optimization (Phase Ib): 2 or 3 doses & schedule selected from Part 1: From the lower limit [Optimal Biologically Active Dose (OBD)] & upper limit [Maximum Tolerated Dose (MTD) or Maximum Administered Dose (MAD) if MTD is not reached]
  Part 3: Dose Expansion at RP2D (Phase II): To be defined later on
  Interventions: Drug: VERT-002

INTERVENTIONS:
Drug: VERT-002 — Route of Administration: Intravenous
  Other Names: PFL-002

SUMMARY:
The goal of this clinical trial is to investigate the safety, the activity of VERT-002 (PFL-002), and the optimal safe dose to be used, in participants with solid tumors including non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Part 1: histological confirmation of relapsed and/or refractory locally advanced or metastatic solid tumor for which no standard of care treatment is available.
2. Part 2: histological confirmation of locally advanced or metastatic NSCLC Stage IIIB/C or IV (American Joint Commission on Cancer [AJCC] 8th edition) in participants who are not eligible for or should have received available standard of care therapies including curative intent surgery, chemoradiation, radiotherapy or systemic therapy.
3. Part 1: presence of at least one of the following MET alterations based on local documentation of blood or archived tissue results:

   * METex14 mutation
   * MET kinase domain activating gene mutations (e.g. H1094L/R/Y, D1228H/N/V, Y1230A/C/D/H)
   * MET amplification
4. Part 2-a: presence of METex14 mutation (based on local documentation of blood or archived tissue results) and for Part 2-b presence of at least one of the following MET alterations: METex14 mutation (based on local documentation of blood or archived tissue results), de novo MET amplification (based on local documentation of archived tissue results). Confirmation after enrollment in the trial will be performed by central testing from an archival tumor biopsy sample (either tissue block or at least 15 serial cut unstained slides of 5 μm, at least 20% tumor content). In case no archival biopsy is available for central testing, the patient must be willing to have a fresh tumor biopsy sample collected and the tumor biopsy should be deemed safe and feasible by the investigator.
5. Part 2: at least one measurable target lesion according to RECIST v1.1.
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
7. Part 1: participants may have received MET Tyrosine Kinase Inhibitor (TKI) as part of previous treatment, regardless of the line of therapy (first or second line), and regardless of the MET TKI being combined or not. Note: crizotinib will be considered a MET TKI.
8. Part 2: a maximum of 3 prior lines of systemic therapies.
9. Adequate hematologic function.
10. Adequate hepatic function.
11. Adequate renal function.
12. Albumin ≥ 3 g/dL.
13. Adequate coagulation function.
14. Adequate cardiac function.
15. Female participants of childbearing potential must have a negative highly sensitive serum β-HCG test performed within 7 days prior to the first dose of VERT-002 and a negative urine pregnancy test performed at C1D1 prior to the first dose of VERT-002.
16. Male participants/partners with female spouse/partners of childbearing potential must agree to take appropriate precautions to avoid fathering a child.

NOTE: Other protocol defined inclusion criteria may apply.

Exclusion Criteria:

1. Part 2: Documented evidence by local testing of targetable oncogene driver mutations.
2. History of a primary malignancy other than the cancer under trial (as defined for Parts 1 and 2) with the exception of:

   * Participants with a previous malignancy who completed their anticancer treatment at least 2 years before signing informed consent and with no evidence of residual disease from the prior malignancy at screening.
   * Malignancies with a negligible risk of metastasis or death (i.e. 5-year overall survival rate > 90%) that are adequately treated.
3. Uncontrolled Central Nervous System (CNS) metastases or spinal cord compression that are associated with progressive neurological symptoms or require increasing doses of corticosteroids to control the CNS disease.
4. History of hypersensitivity to active or inactive ingredients of VERT-002, or drugs with a similar chemical structure or from a similar class.
5. Active, bacterial, fungal, or viral infection, within 2 weeks prior to the first dose of VERT-002 (C1D1).
6. Positive SARs-CoV-2 or variants of SARs-CoV2 test within 2 weeks prior to first dose administration of VERT-002 (C1D1) or with suspected infection with SARs-CoV-2 or variants of SARs-CoV-2 and confirmation pending.
7. Impaired cardiovascular function or clinically significant cardiovascular disease (either active or within 6 months prior to signing main informed consent).
8. Uncontrolled intercurrent illness including, but not limited to psychiatric illness or social situation that would limit compliance with trial requirements.
9. Past medical history of Interstitial Lung Disease (ILD), drug induced ILD, radiation pneumonitis that requires steroid treatment, or any evidence of clinically active ILD.
10. Women who are pregnant or breastfeeding.
11. Prior anticancer therapy:

    * MET TKI within 7 days prior to the first dose of VERT-002,
    * Any other systemic anticancer therapy within 28 days or 5 half-lives of the anticancer therapy whichever is the shortest, but with a minimum of 14 days interval, prior to the first dose of VERT-002 (C1D1),
    * Radiotherapy to a large field or including a vital organ (including whole brain radiotherapy or stereotactic radiosurgery to brain) within 14 days prior to the first dose of VERT-002 (C1D1).
12. Live attenuated vaccine within 28 days prior to the first dose of VERT-002 (C1D1).
13. Any toxicities from prior therapy with NCI- CTCAE Grade > 1 at the time of the first dose administration of VERT-002 (C1D1). Exceptions include any grade alopecia, fatigue and peripheral neuropathy with a grade ≤ 2.
14. Major surgical procedure within 14 days of the first dose of VERT-002 (C1D1).
15. Participation in a clinical trial with administration of an investigational drug within 5 half- lives plus 14 days of the investigational drug, prior to the first dose of VERT-002 (C1D1).

NOTE: Other protocol defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2030-10-21 (Estimated); Study Completion 2032-10-01 (Estimated)

PRIMARY OUTCOMES:
Safety: All parts: Incidence and severity of treatment emergent adverse events (TEAEs)/serious adverse events (SAEs), according to NCI-CTCAE v5.0 criteria. | Screening to Safety Follow-up (30 days post last dose)
Tolerability: All parts: Incidence of TEAEs/SAEs leading to VERT-002 dose reduction, interruption or discontinuation. | From screening up to 13 months
Part 1: Maximum Tolerated Dose (MTD): Incidence of Dose-Limiting Toxicities (DLTs) | From the start of trial treatment until end of Cycle 1 per dose level
Part 1: Optimal Biologically Active Dose (OBD): Incidence on PK/PD and ORR (Objective Response Rate) | From the first VERT-002 intake up to 13 months
Part2a: Preliminary activity assessment: ORR and cORR (Confirmed Objective Response Rate) | From the start of trial treatment up to 13 months
Part2b: Recommended Phase 2 Dose (RP2D): Incidence on overall safety, PK, PDs and cORR | From the start of trial treatment up to 13 months

SECONDARY OUTCOMES:
Serum PK Parameter: Maximum Plasma Concentration (Cmax) | Part 1: Cycle 1 and Cycle 2 - Days 1,2,4,8,15 and 22; Cycle 3 onward Day 1 and EOT (up to 8 months). Part 2: Cycle 1 Days 1,8 and 15; Cycle 2 Days 1 and 15; Cycle 3 onward Day 1; and EOT (up to 12 months). Each cycle is 28 Days
Serum PK Parameter: PK exposure parameter: Area Under The Plasma Concentration-Time Curve From Time Zero To Dosing Interval (AUC0-tau) | Part 1: Cycle 1 and Cycle 2 - Days 1,2,4,8,15 and 22; Cycle 3 onward Day 1 and EOT (up to 8 months). Part 2: Cycle 1 Days 1,8 and 15; Cycle 2 Days 1 and 15; Cycle 3 onward Day 1; and EOT (up to 12 months). Each cycle is 28 Days
Serum PK Parameter: Accumulation Ratio (Rac) for Maximum Observed Concentration (Cmax) and Area Under The Concentration-Time Curve (AUC) | Part 1: Cycle 1 and Cycle 2 - Days 1,2,4,8,15 and 22; Cycle 3 onward Day 1 and EOT (up to 8 months). Part 2: Cycle 1 Days 1,8 and 15; Cycle 2 Days 1 and 15; Cycle 3 onward Day 1; and EOT (up to 12 months). Each cycle is 28 Days
Serum PK Parameter: Trough Concentration (Ctrough) | Part 1: Cycle 1 and Cycle 2 - Days 1,2,4,8,15 and 22; Cycle 3 onward Day 1 and EOT (up to 8 months). Part 2: Cycle 1 Days 1,8 and 15; Cycle 2 Days 1 and 15; Cycle 3 onward Day 1; and EOT (up to 12 months). Each cycle is 28 Days
Serum ADA Parameter: Incidence of VERT-002 anti- drug antibodies (ADA) | Parts 1 and 2: Cycle 1 Days 1,8, and 15; Cycle 2 Days 1 and 15; Cycle 3 onward Day 1; and EOT (up to 8 months). Each cycle is 28 Days
All Parts: cORR (Confirmed Objective Response Rate) based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 per Investigator's Reviewer (IR) | From the start of the treatment to at least 80% of the participants have been followed up for 24 months
All Parts: DCR (Disease Control Rate) based on RECIST version 1.1 per IR | From the start of the treatment to at least 80% of the participants have been followed up for 24 months
All Parts: TTR (Time To Response) according to RECIST version 1.1 per IR | From the start of the treatment to at least 80% of the participants have been followed up for 24 months
All Parts: Duration Of Response (DOR) according to RECIST v1.1 per IR | From the start of the treatment to at least 80% of the participants have been followed up for 24 months
Part 2: Progression Free Survival (PFS) according to RECIST v1.1 per IR | From the start of the treatment to at least 80% of the participants have been followed up for 24 months
Part 2: Overall Survival (OS) | From the start of the treatment to at least 80% of the participants have been followed up for 24 months

CONTACTS AND LOCATIONS:
Locations (19):
- United States (3):
  - Georgetown Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - Gabrail Cancer Research Center, Canton, Ohio
  - Sarah Cannon Research Institute Oncology Partners, Nashville, Tennessee
- Institut Jules Bordet, Anderlecht, Belgium
- France (4):
  - APHP de Marseille - Hôpital Nord, Marseille
  - Institut de Cancerologie de Ouest (ICO) - Saint-Herblain, Saint-Herblain
  - Institut Universitaire du Cancer de Toulouse - Oncopole, Toulouse
  - Gustave Roussy, Villejuif
- Germany (2):
  - Universitaet zu Koeln - Centrum fuer Integrierte Onkologie (CIO), Cologne
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
- Azienda Ospedaliero - Universitaria San Luigi Gonzaga, Orbassano, Italy
- Nederlands Kanker Instituut - Antoni van Leeuwenhoek Ziekenhuis, Amsterdam, Netherlands
- South Korea (2):
  - Yonsei University College of Medicine, Seoul
  - Asan Medical Center (AMC), Seoul
- Spain (2):
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
- Taiwan (3):
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Pierre Fabre is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies as defined in our commitments. These requests are reviewed and approved by an independent review panel on the basis of scientific ground. All data provided if any is anonymized to respect the privacy of trial participants in line with applicable laws and regulations.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: This trial data availability is according to the criteria and process described on our website.

REFERENCES:
- See also: For eligible studies, qualified researchers may request access to individual patient level clinical data. See Pierre Fabre's commitment to transparency of clinical study information Pillar 5. — https://clinicaltrials.pierre-fabre.com/en/our-commitments